CLINICAL TRIAL: NCT06726057
Title: A Multi-component Intervention for Controlling Hypertension in the Adult Rural Population of Pakistan: a Protocol for a Hybrid Type III Implementation-effectiveness Cluster Randomized Controlled Trial
Brief Title: Implementing a Multi-component Hypertension Control Strategy in Rural Pakistan
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: University of York (Other)
Responsible Party: Principal Investigator, Zainab Samad, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-9084-26739
Record Dates: First submitted 2024-10-29; First posted 2024-12-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: multicomponent hypertension intervention; rural PAkistan; primary care setting; basic health unit; lady health workers; community health workers; hypertension in rural adult population; health education; blood pressure monitoring by community health workers; referrals; hypertension management; implementation trial; hybrid type III trial; implementation effectiveness trial; cluster randomized controlled trial; trial on hypertension; CFIR; ERIC; consolidated framework for implementation research; expert recommendations for implementation change; general practitioners; doctors; control of blood pressure; community based intervention for control of hypertension
MeSH Terms: conditions — Hypertension; Health Education

STUDY DESIGN:
Intervention Model Description: Hybrid type III implementation-effectiveness cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent hypertension intervention (Active Comparator): The multicomponent hypertension intervention arm (control arm) will receive the proven multicomponent hypertension intervention (MCHI) comprising four components.
  Interventions: Behavioral: Multicomponent hypertension intervention
- Implementation strategies in conjunction with multicomponent hypertension intervention (Experimental): Implementation strategies in conjunction with multicomponent hypertension intervention arm (Intervention arm) will receive implementation strategies in conjunction with multi-component hypertension intervention (MCHI)
  Interventions: Behavioral: Imlementation strategies in conjunction with multicomponent hypertension intervention

INTERVENTIONS:
Behavioral: Imlementation strategies in conjunction with multicomponent hypertension intervention — In this study, the researchers will develop and test strategies for the implementation and scale-up of a proven multicomponent hypertension intervention (MCHI) programme in Pakistan. Implementation strategies will be devised through an engagement process and will involve the use of implementation frameworks including the Consolidated Framework for Implementation Research (CFIR) to identify barriers and facilitators to the implementation of MCHI& Expert Recommendations for Implementation Change (ERIC) to identify a set of implementation strategies addressing each barrier. Input for the development of strategies will be sought from the community, public health sector managers, general practitioners and community health workers. The implementation strategies will be used to randomise study clusters while MCHI will be implemented in both intervention and control arms.
  Arms: Implementation strategies in conjunction with multicomponent hypertension intervention
Behavioral: Multicomponent hypertension intervention — The multicomponent hypertension intervention has four components as follows:
  1. Training of community health workers (CHWs) in conducting health education sessions regarding hypertension, its risk factors, prevention, and health-seeking
  2. Blood pressure (BP) monitoring and referral of hypertensive individuals by CHWs to general practitioners in primary care facilities
  3. Training of general practitioners in primary care settings in BP monitoring and management of hypertension
  4. Hypertension care coordination in primary care facilities for the care of referred patients.
  Arms: Multicomponent hypertension intervention

SUMMARY:
This is a research about cardiovascular disease risk reduction: a comprehensive package for the reduction of risk in Sindh, Pakistan. The research is being conducted by the Aga Khan University and is funded by the National Institute of Health and Care Research UK.

Hypertension is a major public health concern globally. It is a significant risk for cardiovascular disease (CVD) and premature death. In Pakistan, the prevalence of hypertension, including those on medication, is high. However, there are also high rates of undertreatment and underdiagnosis of hypertension in Pakistan. Addressing the prevention and control of CVD requires a multi-faceted approach that targets diverse populations across different settings. In some populations, we have interventions that have been proven effective but have not been implemented for example in rural communities. In Pakistan, prior community-based trial regarding multi-component hypertension intervention has proven to be effective in reducing blood pressure. However, the findings of this work have not translated to change in practice on the ground suggesting the need for implementation research to examine the best ways to implement this intervention in the real world. Hence, in this study researchers aim to assess the impact of this evidence-based intervention when implemented at scale in rural communities.

Participants will be asked to participate in a research study designed to improve their blood pressure control. This study enrols participants aged 35 years and above. As part of this study, they will undergo:

* blood pressure measurements at regular intervals by lady health workers
* home health education sessions conducted by lady health workers
* participants may be referred to a nearby health facility/qualified medical practitioners for management of high blood pressure
* baseline survey at the start of the study having questions about participants' medical history, risk factors for cardiovascular disease and high blood pressure and bodily measurements including weight, height and waist circumference
* follow-up surveys every 6 months for 2 years. The survey questions will comprise of medical history, risk factors for cardiovascular disease and high blood pressure; and bodily measurements including weight, height and waist circumference
* blood and urine samples for testing at baseline survey and during endline survey

POSSIBLE RISKS OR DISCOMFORT

There are no risks involved as a result of participants' participation in this study except for their time. Since they will be followed up for 2 years, any new information developed during the study that may affect their willingness to continue participation will be communicated to them. Participants may feel a little discomfort at the site of the needle prick when drawing a blood sample.

POSSIBLE BENEFITS

Participants will be able to know about their risk of high blood pressure and cardiovascular disease. They'll be referred to a qualified medical practitioner for the management of your high blood pressure. Also, the results of their blood and urine tests will be shared with participants that will help them know about their health.

The main contact for this research study is the principal investigator Dr Zainab Samad (02134864660).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥35 years
2. Residents of the selected clusters
3. Have hypertension defined as either:

   * Persistently elevated BP (Systolic blood pressure [SBP] SBP ≥140 mm Hg or diastolic blood pressure [DBP] DBP ≥90 mm Hg) from each set of the last two of the three readings from two separate days, where BP measurements on the same day were measured at least 1 minute apart OR
   * Diagnosed previously by a physician as hypertensive and/or on antihypertensive medications.

Exclusion Criteria:

1. Pregnant women and persons with advanced illness (e.g., those receiving dialysis or with liver failure), cancer
2. Unable to travel to the clinic
3. Unwilling/unable to provide consent

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3476 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
BP-lowering medications per participant | From enrollment to the end of Intervention at 24 months
  After estimating the proportional change in the number between the baseline and the 24-month follow-up, the mean difference between both the study arms will be estimated. A mean difference of 0.1 would be considered clinically significant.

OTHER OUTCOMES:
Implementation outcomes [as per RE-AIM framework domain of Adoption ] | From enrollment to the first 12 months of Intervention
  The proportion of LHWs from 30 study clusters conducting HHE sessions, monitoring blood pressure and doing referrals of hypertensive patients to health facilities during the first 12 months Data source: HHE and referral checklists by LHWs, Baseline/follow-up survey
Implementation outcomes [as per RE-AIM framework domain of Adoption ] | From enrollment to the first 12 months of Intervention
  The proportion of GPs from 30 study clusters screening and providing hypertension management to hypertensive patients at BHU/RHC referred by LHW during the first 12 months Data source: GP checklists, Baseline/follow-up surveys
Implementation outcomes [as per RE-AIM framework domain of Implementation] | From enrollment to the end of Intervention at 24 months
  The mean number of the planned home visits/participant over 24 months (a maximum of sixteen visits, one every 3 months, are planned per participant) by LHW for HHE and BP monitoring Data source: LHWs' HHE and referral checklists, Baseline/follow-up surveys
Implementation outcomes [as per RE-AIM framework domain of Implementation] | From enrollment to the end of Intervention at 24 months
  The mean number of healthcare contacts with GPs at the Basic Health Unit per participant over 24 months among those identified as having uncontrolled BP (SBP≥140 mm Hg and/or DBP≥90 mm Hg) by LHW at one or more than one occasion during the trial Data source: GP checklists, Baseline/follow-up surveys
Implementation outcomes [as per RE-AIM framework domain of Maintenance] | From enrollment to the end of Intervention at 24 months
  The proportion of participants receiving visits by LHWs for HHE and BP monitoring at 6, 12, and 24 months.
  Data source: LHWs' HHE & referral checklists, Baseline/follow-up surveys
Implementation outcomes [as per RE-AIM framework domain of Maintenance] | From enrollment to the end of Intervention at 24 months
  The proportion of participants that received advice and/or treatment from the GPs at the Basic Health Unit after being identified as having uncontrolled BP (SBP≥140 mm Hg and/or DBP≥90 mm Hg) by LHW at 6, 12, and 24 months.
  Data source: GP checklists, Baseline/follow-up surveys
Effectiveness outcomes | From enrollment to the end of Intervention at 24 months
  Health-related quality of life i.e., EQ-5D-5L range, 0 to 100, with higher scores indicating better health.
Effectiveness outcomes | From enrollment to the end of Intervention at 24 months
  The proportion of participants with blood-pressure control (SBP 140 mmHg and DBP 90 mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith JD, Hasan M. Quantitative approaches for the evaluation of implementation research studies. Psychiatry Res. 2020 Jan;283:112521. doi: 10.1016/j.psychres.2019.112521. Epub 2019 Aug 17. PMID 31473029
- [Background] Riaz M, Shah G, Asif M, Shah A, Adhikari K, Abu-Shaheen A. Factors associated with hypertension in Pakistan: A systematic review and meta-analysis. PLoS One. 2021 Jan 29;16(1):e0246085. doi: 10.1371/journal.pone.0246085. eCollection 2021. PMID 33513161
- [Background] Turana Y, Tengkawan J, Chia YC, Nathaniel M, Wang JG, Sukonthasarn A, Chen CH, Minh HV, Buranakitjaroen P, Shin J, Siddique S, Nailes JM, Park S, Teo BW, Sison J, Ann Soenarta A, Hoshide S, Tay JC, Prasad Sogunuru G, Zhang Y, Verma N, Wang TD, Kario K; HOPE Asia Network. Hypertension and stroke in Asia: A comprehensive review from HOPE Asia. J Clin Hypertens (Greenwich). 2021 Mar;23(3):513-521. doi: 10.1111/jch.14099. Epub 2020 Nov 15. PMID 33190399
- [Background] Forouzanfar MH, Liu P, Roth GA, Ng M, Biryukov S, Marczak L, Alexander L, Estep K, Hassen Abate K, Akinyemiju TF, Ali R, Alvis-Guzman N, Azzopardi P, Banerjee A, Barnighausen T, Basu A, Bekele T, Bennett DA, Biadgilign S, Catala-Lopez F, Feigin VL, Fernandes JC, Fischer F, Gebru AA, Gona P, Gupta R, Hankey GJ, Jonas JB, Judd SE, Khang YH, Khosravi A, Kim YJ, Kimokoti RW, Kokubo Y, Kolte D, Lopez A, Lotufo PA, Malekzadeh R, Melaku YA, Mensah GA, Misganaw A, Mokdad AH, Moran AE, Nawaz H, Neal B, Ngalesoni FN, Ohkubo T, Pourmalek F, Rafay A, Rai RK, Rojas-Rueda D, Sampson UK, Santos IS, Sawhney M, Schutte AE, Sepanlou SG, Shifa GT, Shiue I, Tedla BA, Thrift AG, Tonelli M, Truelsen T, Tsilimparis N, Ukwaja KN, Uthman OA, Vasankari T, Venketasubramanian N, Vlassov VV, Vos T, Westerman R, Yan LL, Yano Y, Yonemoto N, Zaki ME, Murray CJ. Global Burden of Hypertension and Systolic Blood Pressure of at Least 110 to 115 mm Hg, 1990-2015. JAMA. 2017 Jan 10;317(2):165-182. doi: 10.1001/jama.2016.19043. PMID 28097354
- [Background] Gaglio B, Shoup JA, Glasgow RE. The RE-AIM framework: a systematic review of use over time. Am J Public Health. 2013 Jun;103(6):e38-46. doi: 10.2105/AJPH.2013.301299. Epub 2013 Apr 18. PMID 23597377
- [Background] Powell BJ, Waltz TJ, Chinman MJ, Damschroder LJ, Smith JL, Matthieu MM, Proctor EK, Kirchner JE. A refined compilation of implementation strategies: results from the Expert Recommendations for Implementing Change (ERIC) project. Implement Sci. 2015 Feb 12;10:21. doi: 10.1186/s13012-015-0209-1. PMID 25889199
- [Background] Waltz TJ, Powell BJ, Fernandez ME, Abadie B, Damschroder LJ. Choosing implementation strategies to address contextual barriers: diversity in recommendations and future directions. Implement Sci. 2019 Apr 29;14(1):42. doi: 10.1186/s13012-019-0892-4. PMID 31036028
- [Background] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Wolfenden L, Foy R, Presseau J, Grimshaw JM, Ivers NM, Powell BJ, Taljaard M, Wiggers J, Sutherland R, Nathan N, Williams CM, Kingsland M, Milat A, Hodder RK, Yoong SL. Designing and undertaking randomised implementation trials: guide for researchers. BMJ. 2021 Jan 18;372:m3721. doi: 10.1136/bmj.m3721. PMID 33461967
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Ostermann J, Brown DS, de Bekker-Grob EW, Muhlbacher AC, Reed SD. Preferences for Health Interventions: Improving Uptake, Adherence, and Efficiency. Patient. 2017 Aug;10(4):511-514. doi: 10.1007/s40271-017-0251-y. No abstract available. PMID 28597375
- [Background] Heerden A, Ntinga X, Lippman SA, Leslie HH, Steward WT. Understanding the Factors that Impact Effective Uptake and Integration of Health Programs in South African Primary Health Care Clinics. Res Sq [Preprint]. 2021 Aug 17:rs.3.rs-783631. doi: 10.21203/rs.3.rs-783631/v1. PMID 34426806
- [Background] Schwalm JR, McCready T, Lamelas P, Musa H, Lopez-Jaramillo P, Yusoff K, McKee M, Camacho PA, Lopez-Lopez J, Majid F, Thabane L, Islam S, Yusuf S. Rationale and design of a cluster randomized trial of a multifaceted intervention in people with hypertension: The Heart Outcomes Prevention and Evaluation 4 (HOPE-4) Study. Am Heart J. 2018 Sep;203:57-66. doi: 10.1016/j.ahj.2018.06.004. Epub 2018 Jun 22. PMID 30015069
- [Background] Jafar TH, Gandhi M, de Silva HA, Jehan I, Naheed A, Finkelstein EA, Turner EL, Morisky D, Kasturiratne A, Khan AH, Clemens JD, Ebrahim S, Assam PN, Feng L; COBRA-BPS Study Group. A Community-Based Intervention for Managing Hypertension in Rural South Asia. N Engl J Med. 2020 Feb 20;382(8):717-726. doi: 10.1056/NEJMoa1911965. PMID 32074419
- [Background] Elahi A, Ali AA, Khan AH, Samad Z, Shahab H, Aziz N, Almas A. Challenges of managing hypertension in Pakistan - a review. Clin Hypertens. 2023 Jun 15;29(1):17. doi: 10.1186/s40885-023-00245-6. PMID 37316940
- [Background] Rafique I, Saqib MAN, Munir MA, Qureshi H, Rizwanullah, Khan SA, Fouad H. Prevalence of risk factors for noncommunicable diseases in adults: key findings from the Pakistan STEPS survey. East Mediterr Health J. 2018 Apr 5;24(1):33-41. PMID 29658619
- [Background] Basit A, Tanveer S, Fawwad A, Naeem N; NDSP Members. Prevalence and contributing risk factors for hypertension in urban and rural areas of Pakistan; a study from second National Diabetes Survey of Pakistan (NDSP) 2016-2017. Clin Exp Hypertens. 2020;42(3):218-224. doi: 10.1080/10641963.2019.1619753. Epub 2019 May 31. PMID 31151358
- [Background] Gaziano TAJPHACDPM: Cardiovascular diseases worldwide. 2022, 1:8-18.
- [Background] Mendis S, Graham I, Narula J. Addressing the Global Burden of Cardiovascular Diseases; Need for Scalable and Sustainable Frameworks. Glob Heart. 2022 Jul 29;17(1):48. doi: 10.5334/gh.1139. eCollection 2022. PMID 36051329
- [Background] Hu B, Shi Y, Zhang P, Fan Y, Feng J, Hou L. Global, regional, and national burdens of hypertensive heart disease from 1990 to 2019 ：A multilevel analysis based on the global burden of Disease Study 2019. Heliyon. 2023 Nov 23;9(12):e22671. doi: 10.1016/j.heliyon.2023.e22671. eCollection 2023 Dec. PMID 38213586
- [Derived] Naeem I, Almas A, Sheikh A, Hewitt C, Khwaja H, Afaq S, Bukhari S, Soofi S, S Virani S, Hanif S, Hashmi S, Walker S, Bhutta ZA, Siddiqi K, Samad Z. Multicomponent intervention for controlling hypertension in the adult rural population of Pakistan: a protocol for a hybrid type III implementation-effectiveness cluster randomised controlled trial. BMJ Open. 2025 Jun 27;15(6):e100365. doi: 10.1136/bmjopen-2025-100365. PMID 40578881
- See also: Provisional summary results of 6th population and housing census-2017. Matiari district — https://www.pbs.gov.pk/census-2017-district-wise/results/087
- See also: Updated CFIR Constructs — https://cfirguide.org/evaluation-design/overview/
- See also: Use of Iterative PRISM and RE-AIM During Implementation — https://re-aim.org/applying-the-re-aim-framework/re-aim-guidance/use-during-implementation/

DOCUMENTS (8):
  • Study Protocol and Statistical Analysis Plan: 5. CVD Study Protocol V5 08112025 CT 1.4 (2025-11-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: CVD Study Protocol V1.2 (2025-04-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: CVD Study Protocol V1.1 (2024-10-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: CVD Study Protocol V1.3 (2025-08-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/Prot_SAP_003.pdf
  • Study Protocol and Statistical Analysis Plan: 6. CVD Study Protocol V6 27012026 (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/Prot_SAP_007.pdf
  • Informed Consent Form: Informed consent baseline recruitment (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/ICF_004.pdf
  • Informed Consent Form: Informed consent workshop participants (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/ICF_005.pdf
  • Informed Consent Form: Informed consent Screening (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT06726057/ICF_006.pdf